CLINICAL TRIAL: NCT01400633
Title: A Prospective Multicenter Observational Study for Dacogen Long-Term Treatment in Patients With Myelodysplastic Syndrome
Brief Title: An Observational Study for Dacogen Long-Term Treatment in Patients With Myelodysplastic Syndrome
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR017842; DACOGENMDS4013 (Other: Janssen Korea, Ltd., Korea); Long-term treatment of Dacogen (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2011-07-14; First posted 2011-07-22 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic Syndrome; Dacogen; decitabine; epigenetic therapy; hypomethylating agent
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Decitabine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 001: decitabine injection decitabine intravenous injection 20mg/m2 once a day for 5 consecutive days every 4 weeks
  Interventions: Drug: decitabine injection

INTERVENTIONS:
Drug: decitabine injection — decitabine intravenous injection 20mg/m2 once a day for 5 consecutive days every 4 weeks

SUMMARY:
The purpose of this study is to investigate the overall response rate (ORR) and safety when treating patients with myelodysplastic syndrome with decitabine. Decitabine is to be administered as long as there is evidence of clinical benefit.

DETAILED DESCRIPTION:
This study is a prospective (the study follows a group of individuals over time), open label (all people involved know the identity of the intervention), multicenter, single arm (one group of patients receiving the same treatment), observational study to observe the response rate and safety of decitabine when treating patients with myelodysplastic syndrome with decitabine. Decitabine is to be administered as long as there is evidence of clinical benefit. It will be assessed if the treatment duration could be prolonged by appropriate toxicity management such as an active antibiotic prophylaxis or dose and schedule modification, and whether this leads to potentially increased clinical benefits such as higher response rate, longer time to Acute Myeloid Leukemia, and prolonged overall survival. For safety evaluation, adverse events and peripheral blood findings will be collected. The patient will receive decitabine intravenous injection 20mg/m2 once a day for 5 consecutive days every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with (primary or secondary) Myelodysplastic Syndrome including Chronic Myelomonocytic Leukemia (CMML)
* Patients with an International Prognostic Scoring System >= Int-1
* Patients who were never treated with hypomethylating agent (azacitidine and decitabine)
* Female patients who are postmenopausal or received contraceptive operation or refrain from sexual relations. Women of childbearing potential should conduct an effective method of birth control (oral contraceptives, injections, intrauterine device, double barrier method, contraceptive patch and male partner's sterilization), in case of male patients who will not have a baby within 2 months after the completion of decitabine therapy
* Patients who signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study.

Exclusion Criteria:

* Patients diagnosed with Acute Myelogenous Leukemia (AML, bone marrow stem cell counts exceeding 20%) or other progressive malignant diseases
* Patients with active infection of virus or bacteria
* Patients who used to be treated with azacitidine or decitabine
* Patients who are hypersensitive to excipients of decitabine
* Patients who are pregnant or breast-feeding.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Secondary or tertiary hospitals in South Korea
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2010-12; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
overall response rate | every 28 days up to approximately 5 years

SECONDARY OUTCOMES:
The change of transfusion requirements | every 4 weeks up to approximately 5 years
Overall survival | every 3 months up to approximately 5 years
Adverse events | every 4 weeks up to approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd. Clinical Trial, Study Director — Janssen Korea, Ltd.
Locations (16):
- South Korea (16):
  - Ansan
  - Anyang
  - Busan
  - Cheonan
  - Chungcheongbuk-Do
  - Daegu
  - Daejeon
  - Gyeonggi-do
  - Hwasun Gun
  - Incheon
  - Jinju
  - Jungnam
  - Kwanju
  - Pusan
  - Seoul
  - Suwon

REFERENCES:
- [Derived] Jung KS, Kim YJ, Kim YK, Park SK, Kim HG, Kim SJ, Park J, Choi CW, Do YR, Kim I, Park S, Mun YC, Jeong SH, Kim MK, Yi HG, Chang MH, Kim SY, Lee JH, Jang JH. Clinical Outcomes of Decitabine Treatment for Patients With Lower-Risk Myelodysplastic Syndrome on the Basis of the International Prognostic Scoring System. Clin Lymphoma Myeloma Leuk. 2019 Oct;19(10):656-664. doi: 10.1016/j.clml.2019.06.003. Epub 2019 Jun 27. PMID 31375393